CLINICAL TRIAL: NCT01511679
Title: Brain-imaging and Adolescent Neuroscience Consortium
Acronym: BANC
Status: Withdrawn | Type: Observational
Why Stopped: The project was not funded.
Sponsor: Boston Children's Hospital (Other)
Collaborators: Massachusetts General Hospital (Other); Mclean Hospital (Other); Massachusetts Institute of Technology (Other)
Responsible Party: Sponsor
Other Study IDs: BANC RFA-AA-12-006
Record Dates: First submitted 2012-01-13; First posted 2012-01-19 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2013-01

CONDITIONS: Alcohol Abuse
Keywords: Alcohol abuse
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva DNA samples for future analyses.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Alcohol-naive adolescents: A general population longitudinal cohort of alcohol-naïve (or h/o minimal recent-onset drinking) adolescents in three specific age-groups: early (12-14 y/o), middle (15-17 y/o), and late (18-21 y/o).
- Treatment sample: A sample of adolescents who have a >1 year history of heavy drinking but have agreed to stop drinking as part of their treatment plan
- High risk sample: High-risk adolescents who have a family history of alcohol-use disorder and other risk factors (symptoms of Attention-Deficit/Hyperactivity Disorder (ADHD), Conduct Disorder, or Mood Disorder)

SUMMARY:
This is a multi-site study of adolescents 12-21 years-of-age to evaluate the long and shorter-term effect of adolescent alcohol use on the developing brain.

DETAILED DESCRIPTION:
The overall specific aims of this study are to: 1) assess the short and long-term consequences of alcohol exposure on brain, cognitive, and emotional/regulatory development during preadolescence and adolescence; 2) determine the effects of timing, dose, and duration of alcohol on brain and cognitive development; 3) assess recovery of neural and behavioral function to determine if the plasticity of the adolescent brain makes it more or less vulnerable to alcohol's acute and chronic effects; 4) understand how other key covariates (e.g., existing or emerging psychopathology, family history of alcoholism, demographics, pubertal development) factor into alcohol's effects on the brain; and 5) identify early neural, cognitive, and affective markers that may predict alcohol abuse and dependence during adolescence and/or adulthood.

ELIGIBILITY:
Inclusion Criteria:

* able to read and understand English
* available for follow-up
* parental consent/adolescent assent for those 12-17 years
* consent for those 18-21 years

Exclusion Criteria:

* Weight > 300 lbs
* braces or unremovable embedded metal
* claustrophobia or inability to lie still in MRI machine
* current or past 12-mos pregnancy (females)
* requires urgent medical/mental health care

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Male and female adolescents 12-21 years-of-age presenting for care at one of the participating medical clinics
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2017-03 (Estimated); Study Completion 2017-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: John R Knight, MD, Principal Investigator — Boston Children's Hospital; Gordon J Harris, PhD, Principal Investigator — Massachusetts General Hospital; Simon Warfield, PhD, Principal Investigator — Boston Children's Hospital; Avram Holmes, PhD, Principal Investigator — Harvard University; Scott Lukas, PhD, Principal Investigator — Mclean Hospital; Marisa Silveri, PhD, Principal Investigator — Mclean Hospital; Marlene Oscar Berman, PhD, Principal Investigator — Boston University; John Gabrieli, PhD, Principal Investigator — Massachusetts Institute of Technology
Locations (4):
- United States (4):
  - McLean Hospital, Belmont, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston University School of Medicine, Boston, Massachusetts
  - Massachusetts Institute of Technology, Cambridge, Massachusetts

REFERENCES:
- See also: Center for Adolescent Substance Abuse Research at Children's Hospital Boston — http://www.ceasar.org